CLINICAL TRIAL: NCT07403955
Title: A Randomized Controlled Clinical Study on the Effect of Dapagliflozin on Myocardial Strain in Patients With Acute Heart Failure
Brief Title: The Effect of Dapagliflozin on Myocardial Strain in Patients With Acute Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202505-110-2
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Congestive Heart Failure Acute
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Standard treatment combined with dapagliflozin tablet 10mg qd for 3 months
  Interventions: Drug: Dapagliflozin 10mg Tab
- control group (No Intervention): Dapagliflozin tablet 10mg qd was added for two months after one month of standard treatment

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Compared with the control group, dapagliflozin is started within the first month after the onset of acute heart failure.
  Other Names: Standard Treatment
  Arms: intervention group

SUMMARY:
The goal of this clinical trial is to assess the impact of dapagliflozin on myocardial strain in patients with acute heart failure using speckle tracking echocardiography (STE).

The main questions it aims to answer are:

* Does dapagliflozin improve left ventricular remodeling as well as cardiac systolic and diastolic function?
* Can STE more accurately assess the impact of dapagliflozin on myocardial strain in patients with acute heart failure? Researchers will compare patients receiving oral dapagliflozin to those not receiving it to see if dapagliflozin works to improve left ventricular remodeling as well as cardiac systolic and diastolic function.

Participants will:

* Take dapagliflozin or not every day for 1 month
* Take dapagliflozin for the next 2 months
* Visit the clinic at Month 1 and Month 3 for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from patient or next of kin； Eighteen years and older; Admitted to hospital due to acute heart failure； eGFR> 25ml /min/1.73m2 (calculated by the MDRD equation)； Eligible patients will be enrolled within 24 hours to 14 days after admission, while still hospitalized and in a stable condition.

Exclusion Criteria:

* Type I diabetes mellitus; Systolic blood pressure < 90mmHg at enrollment or positive inotropic drugs are required at enrollment or are expected to be used during hospitalization; Non-cardiac dyspnea； Known hypersensitivity to dapagliflozin； Previous treatment with any SGLT2 inhibitor； History of diabetic ketoacidosis within 3 months； Patients on dialysis； Current atrial fibrillation； Poor echocardiographic images quality prohibiting speckle tracking echocardiography analysis； History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3) or asymptomatic sustained ventricular tachycardia，congenital long QT syndrome, history of QT prolongation associated with other medications that required discontinuation of that medication; Diagnosis of hypertrophic obstructive cardiomyopathy, reversible cardiomyopathy (such as stress cardiomyopathy), cardiac infiltrative diseases (such as myocardial amyloidosis), constrictive pericarditis, severe valvular heart disease (moderate or severe aortic stenosis, severe aortic regurgitation, moderate or severe mitral stenosis, severe mitral regurgitation, heart valve disease expected to undergo surgery during the trial period); Various serious diseases that affect the clinical course of the subjects, such as acute exacerbation of chronic obstructive pulmonary disease and severe liver function impairment (Child-Pugh Grade C), severe anemia (hemoglobin < 90g/L), gastrointestinal surgery or gastrointestinal diseases that may affect the absorption of the test drug, acute or chronic pancreatitis, current urinary or reproductive system infections, and a recorded history of active or suspected malignant tumors or a clear history of malignant tumors within one year prior to screening; Diffuse edema with 4+ edema, estimated blood volume exceeding 40 pounds (18kg); Pregnant, or currently breastfeeding or in the preconception period; Failure to follow the research evaluation schedule for follow-up, or deemed unsuitable for participation by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
left ventricular global longitudinal strain (LVGLS) | at 3 months
  the change in LVGLS from baseline

SECONDARY OUTCOMES:
left ventricular global longitudinal strain (LVGLS) | at 1 month and 3 months
  the change in LVGLS from baseline
peak atrial contraction strain（PACS），peak atrial longitudinal strain（PALS），right ventricular global longitudinal strain（RVGLS） | at 1 month and 3 months
  the change in PACS, PALS, RVGLS from baseline
all-cause mortality， Cardiovascular death， Heart failure hospitalization | at 1 month and 3 months
  The composite secondary endpoint included all-cause mortality, cardiovascular death or heart failure hospitalization

OTHER OUTCOMES:
NYHA functional class, NT-proBNP | at baseline, 1month and 3 months
  NYHA functional class and the level of NT-proBNP

IPD SHARING:
Plan to Share IPD: No